CLINICAL TRIAL: NCT02339857
Title: The Long-term Results of Coronary Artery Bypass Surgery When the No-touch Vein Graft is Anastomised to the Left Anterior Descending Artery.
Brief Title: The Long-term Results of the No-touch Vein Graft to the Left Anterior Descending Artery.
Status: Completed | Type: Observational
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Ninos Samano M.D., Cardiothoracic surgeon, Örebro University, Sweden
Other Study IDs: 102881
Record Dates: First submitted 2015-01-12; First posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Ischemic Heart Disease; Atherosclerosis
Keywords: coronary artery bypass grafting; saphenous vein; grafts
MeSH Terms: conditions — Myocardial Ischemia; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No-touch vein grafts to LAD
  Interventions: Procedure: No-touch harvesting technique

INTERVENTIONS:
Procedure: No-touch harvesting technique — The saphenous vein is harvested with a pedicle of surrounding tissue.

SUMMARY:
The purpose of this study was to investigate whether the no-touch saphenous vein grafts that were used in coronary artery bypass surgery between 2003-2008 had a patency rate comparable to the left internal thoracic artery when the vein grafts were anatomised to the left anterior descending artery.

ELIGIBILITY:
Inclusion Criteria:

1. Coronary artery bypass grafting performed at the Department of Cardiothoracic Surgery, Örebro Universtiy Hospital between 2003-2008.
2. Saphenous vein graft harvesting using the no-touch technique.
3. The saphenous vein anastomised to the left anterior descending artery.
4. Informed consent

Exclusion Criteria:

1. Allergy to contrast media.
2. Impaired renal function.
3. Inability to conduct the study according to protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that performed coronary artery bypass surgery between 2003-2008 and received a no-touch saphenous vein graft to the left anterior descending artery were included consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Total patency of the no-touch vein grafts. | Mean time 8 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ninos Samano, MD, Principal Investigator — Faculty of Medicine and Health, Örebro University, Örebro, Sweden